CLINICAL TRIAL: NCT04343365
Title: Feasibility of Generating Novel Therapeutic Strategies Based on Evolutionary Tumor Board in Cancer Patients
Brief Title: Generating Novel Therapeutic Strategies Based on Evolutionary Tumor Board
Status: Recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-20417
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Incurable Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood collected, and subsequently at designated time points (every 9 weeks from ETB result discussion +/- 4 weeks) depending on the upfront treatment protocol, off therapy, and at disease relapse. For each collection, a total of 20 mL of blood will be drawn, which includes 10 ml of blood in an EDTA tube, and 10 ml in a LBGuard® tube, as described in Lab Manual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants Reviewed by ETB: Participants clinical history, available therapeutic options, and outcome expectations will be presented to the Evolutionary Tumor Board (ETB) along with images and pathology. Strategies and models will be presented regarding additional evolutionary ideas that can be applied.
  Interventions: Other: Evolutionary Tumor Board (ETB)

INTERVENTIONS:
Other: Evolutionary Tumor Board (ETB) — The ETB consists of evolutionary biologists, mathematicians, research scientists, statisticians,data scientists, radiologists, pathologists, oncologists (surgical, radiation, medical, and pediatric), and clinical trial coordinators.The ETB will generate hypotheses, mathematical models, and experiments from the discussion towards further integration of evolutionary ideas towards therapeutic strategies for participants. The ETB will collect data through a chart review regarding adherence and results of ETB recommendation

SUMMARY:
This study will evaluate the ability of a multidisciplinary group, the Evolutionary Tumor Board (ETB), to develop therapeutic strategies in patients without curative options.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be considered likely incurable given a standard of care. This is inclusive of participants in remission but at high risk of recurrence, with suboptimal responses to previous therapy, or with many potentially beneficial, but not curative options for care.
* Participant must have a life expectancy greater than 3 months
* Participant must have an ECOG performance status 0-2
* Participant and primary Oncologist are willing to consider the therapeutic strategies recommended by the ETB
* Willingness to be followed over time and allowing collection of clinical data including scans and serial blood sampling.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who are patients at Moffitt Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
ETB developing therapeutic strategies | Baseline to up to 60 months from end of therapy
  The investigators want to demonstrate the ability of a multidisciplinary group, the ETB, to develop therapeutic strategies in participants without curative options. They plan to enroll 35 patients to this study over 3 years. The primary objective will be successfully met if they can develop an evolutionary based plan that differs from the participants options prior to presentation for at least 80%, or 28 of these participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong Zhang, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided